CLINICAL TRIAL: NCT00914069
Title: Evaluation of the Safety and Effectiveness of the Rapid Intravascular Start (RIVS) System Versus Conventional Catheter for Peripheral Intravenous (PIV) Insertion in Children, Oncology Patients and Elderly: a Controlled Randomized Trial
Brief Title: Effectiveness of the Rapid Intravascular Start (RIVS) System Versus Conventional Catheter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Stopped
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 62009123
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIVS vascular access (Experimental): RIVS vascular access
  Interventions: Device: RIVS vascular access
- Conventional vascular access (Active Comparator): Conventional vascular access
  Interventions: Device: Conventional vascular access

INTERVENTIONS:
Device: RIVS vascular access — Access to peripheral vasculature
  Arms: RIVS vascular access
Device: Conventional vascular access — Vascular access using conventional venous access device
  Arms: Conventional vascular access

SUMMARY:
The study will test a hypothesis that the RIVS system will have a higher rate of successful first PIV placement compared to conventional catheter without a significant increase in complications and time of procedure.

DETAILED DESCRIPTION:
The hypothesis to be statistically tested was that the RIVS system will have a higher rate of successful first attempt peripheral intravenous placement success as compared to conventional peripheral intravenous catheters without a significant increase in device related complications and procedure time.

ELIGIBILITY:
Inclusion Criteria

* Any type of oncology patients undergoing chemotherapy or post-chemotherapy (without a port/cannula), or over 65 years
* Requires peripheral IV as determined by examining physician
* Requires the IV when a study nurse or resident is available
* Able to sign an informed consent

Exclusion Criteria

* Active systemic or cutaneous infection or inflammation;
* Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
* Known, significant history of bleeding diathesis, coagulopathy, von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline International Normalized Ratio (INR) ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
* Currently involved in any other investigational clinical trials;
* Previous vascular grafts or surgery at the target vessel access site;
* Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating;
* Central line available
* Requirement for immediate IV placement (patient's condition would potentially be compromised if there is a time delay in IV placement)

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Stuart, MD, Principal Investigator — Washington Outpatient Surgery Center
Locations (3):
- United States (3):
  - Washington Outpatient Surgery Center, Fremont, California
  - St. Vincent's Medical Center, Jacksonville, Florida
  - University Hospital Case Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to assignment to groups, two subjects withdrew from the study. Also prior to group assignment, one subject did not have a consent form and was excluded from the study.
Period: Overall Study
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Started | 84 | 88
Completed | 84 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIVS Vascular Access | Conventional Vascular Access | Total
Number analyzed (Participants) | 84 | 88 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.4) | 67.2 (10.9) | 66.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data were missing for two (2) subjects.
  Participants
    number analyzed (Participants) | 84 | 86 | 170
    Female | 36 | 49 | 85
    Male | 48 | 37 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 44 | 86
  Black | 10 | 10 | 20
  Asian | 14 | 16 | 30
  Hispanic | 10 | 7 | 17
  Other | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: IV Insertion Success Rate at First Attempt IV Insertion Success Rate at First Attempt
Description: A successful IV insertion includes all of the following: initial vein penetration, which is visualized by a flash back of blood into the access device, deployment of the guidewire, advancement of the catheter into the vein, retraction of needle and guidewire, and flushing of IV. A secured flushed IV will be indicative of a successful PIV placement.
Time Frame: An access attempt usually ranges from 0 to 45 minutes in duration.
Measure: Number; unit: participants
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Number analyzed (Participants) | 84 | 88
participants | 60 | 51
Statistical Analysis 1: Comparison: RIVS Vascular Access vs Conventional Vascular Access; Test type: Superiority or Other; p = 0.05, Fisher Exact — Threshold for significance was p less than or equal to 0.05 by a one-tailed Fisher Exact Test

2. Primary Outcome: Summary of Major Complications
Description: Any device-related or procedure-related adverse event that causes clinically consequential symptoms to the patient. These may include access site hematoma, bleeding, infection, nerve injury, vessel laceration, wound dehiscence, allergic reaction, or inflammation, among others.
Time Frame: Post-PIV placement until catheter removal (usually within 4 days)
Measure: Number; unit: participants
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Number analyzed (Participants) | 84 | 88
participants | 0 | 0

3. Secondary Outcome: Time Required to Obtain Access
Description: A secured flushed IV will be indicative of a successful PIV placement.
Time Frame: An access attempt usually ranges from 0 to 45 minutes in duration.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Number analyzed (Participants) | 84 | 88
minutes | 4.0 (4.0) | 5.0 (5.0)

4. Secondary Outcome: Second Stick Success Rate
Description: A secured flushed IV will be indicative of a successful PIV placement.
Time Frame: An access attempt usually ranges from 0 to 45 minutes in duration.
Population: Number of Participants Analyzed is not consistent with numbers provided in the Participant Flow Module because not all participants required a second attempt at catheter placement.
Measure: Number; unit: participants
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Number analyzed (Participants) | 23 | 36
participants | 10 | 18
Statistical Analysis 1: Comparison: RIVS Vascular Access vs Conventional Vascular Access; Test type: Superiority or Other; p = 0.8, Fisher Exact

5. Secondary Outcome: Summary of Minor Complications
Description: Any device-related or procedure-related adverse event that causes clinically inconsequential symptoms to the patient.
Time Frame: Post-PIV placement until catheter removal (usually within 4 days)
Measure: Number; unit: participants
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Number analyzed (Participants) | 84 | 88
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | RIVS Vascular Access | Conventional Vascular Access
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/88
Other Adverse Events (participants affected / at risk) | 1/84 | 0/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIVS Vascular Access (N=84) | Conventional Vascular Access (N=88)
Minor Vasular Complication (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigators may publish or present the study results with prior consent of the Sponsor, but will not disclose confidential information. Prior to submission by a Principal Investigator for publication or presentation, the Sponsor will be provided with the opportunity to review the submission for confidential information and accuracy.